CLINICAL TRIAL: NCT04325607
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Negative Pressure Wound Therapy With Instillation for Treatment of Hidradenitis Suppurativa
Brief Title: Negative Pressure Wound Therapy With Instillation for Treatment of Hidradenitis Suppurativa
Acronym: HIDRA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was affected by the previous COVID pandemic and patient referral pathway was interrupted
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: KCI Europe Holding B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 247179
Record Dates: First submitted 2020-01-16; First posted 2020-03-27 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Negative pressure wound therapy with instillation; Negative pressure wound therapy
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative Pressure Wound Therapy with instillation (Experimental): Patients in the treatment group will be initiated on VeraFlo instillation (NPWTi) therapy upon excision of HS
  Interventions: Procedure: Excision of HS followed by NPWTi
- Negative Pressure Wound Therapy (Active Comparator): Patient in the control group will be initiated on VAC therapy (NPWT) upon excision of HS
  Interventions: Procedure: Excision of HS followed by NPWT

INTERVENTIONS:
Procedure: Excision of HS followed by NPWTi — The NPWTi that will be used in this study will be the V.A.C. VERAFLO™ Therapy (KCI)
  Other Names: VAC VERAFLO™ Therapy
  Arms: Negative Pressure Wound Therapy with instillation
Procedure: Excision of HS followed by NPWT — The NPWT that will be used in this study will be the V.A.C.® Therapy(KCI)
  Other Names: VAC Therapy
  Arms: Negative Pressure Wound Therapy

SUMMARY:
The current surgical management for severe Hidradenitis suppurativa (HS) involves wide excision of affected skin, resulting in a large soft tissue defect. The soft tissue defect will then be managed with Negative Pressure Wound Therapy (NPWT) to promote healthy granulation tissue formation for wound coverage with Split skin graft (SSG). This long interval between excision and reconstruction could result in long in-patient stay, increased risk of hospital acquired infection and reduced patients' quality of life.

The investigators wish to evaluate the use of Negative Pressure Wound Therapy with instillation (NPWTi), which has potential to allow early wound coverage with SSG, as an alternative to the current standard of care. The investigators hypothesise that NPWTi reduces bacterial load on the wound and allows early wound coverage hence improves patient satisfaction and reduces cost and length of hospital stay.

DETAILED DESCRIPTION:
HS is a recurring chronic skin disease of the hair follicle that usually presents with painful and inflamed lesions in the sweat gland-bearing areas of the body. The lesions often progress to become chronic with pus discharge and scar formation resulting in significant disability.

Current surgical management for severe HS involves surgical removal of all involved hair bearing skin resulting in large areas of soft tissue loss which requires reconstruction. The wound is reconstructed by performing skin grafting, known as SSG, whereby a healthy layer of skin is transferred to the area of tissue loss. SSG enables rapid wound healing and has low risk of recurrence of HS. Skin grafting is often done a few weeks after excision of HS (delayed setting) to ensure higher success rate due to the infected nature of HS. During the interval between surgical removal of areas with HS and skin grafting, the wound is managed with a suction dressing known as the Negative Pressure Wound Therapy (NPWT) to promote formation of healthy wound bed. NPWT is a form of vacuum dressing which applies continuous suction pressure on the wound to remove fluids and bacteria from the wound bed.

The NPWT is highly successful in managing such wounds, however a novel and innovative improvement to this technology with an irrigation system, the Negative Pressure Wound Therapy with instillation (NPWTi), holds promise to enhance production of healthy wound bed and further reducing bacteria and infectious materials from the wound, enabling earlier wound coverage with SSG. The NPWTi involves irrigating and soaking the wound with fluid, followed by removal of the fluid via application of suction pressure at timed, regular intervals. The goal of the instillation therapy is to enable early application of SSG as wound irrigation has long been appreciated as beneficial for cleaning contaminated wounds.

The investigators wish to evaluate the NPWTi as an alternative to NPWT for current surgical management strategy of severe HS. The investigators wish to determine if NPWTi allows early wound coverage with SSG which improves patient satisfaction and reduces length of hospital stay. This research will further our knowledge about the human wound healing process and it may help improve treatment for future patients. The investigators plan to study up to 44 patients in total.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female
2. Age 18-90 at the time of consent
3. Clinical diagnosis of axillary hidradenitis suppurativa
4. Unilateral axillary hidradenitis suppurativa (if bilateral disease, only one side will be included into study).
5. Hidradenitis suppurativa with multiple sinuses which are not able to close directly
6. Not on antibiotics for 6 weeks
7. Patient understands and is willing to participate

Exclusion Criteria:

1. Hidradenitis suppurativa with isolated sinus for direct closure
2. Patient with ongoing chemotherapy or radiotherapy
3. Patient with active cancer
4. Uncontrolled Diabetes Mellitus, as measured by an HbA1c > 10%.
5. BMI over 35
6. Active smoker
7. Presence of one or more medical conditions, including renal, hepatic, hematologic, active auto-immune or immune diseases that, would make the subject an inappropriate candidate for this wound healing study
8. Patient not fit for surgery (ASA classification > 4)
9. Patients not able to consent for procedure in English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
The mean days to wound coverage with split skin graft (SSG) after excision of HS | 2 weeks
  Mean days to wound coverage with split skin graft (SSG) after excision of HS in each treatment arm
The difference in bacterial count on the wound after NPWTi against NPWT | 2 weeks
  Reduction in the number of colony-forming unit (CFU) at each dressing change analysed using tissue culture of wound bed biopsies

SECONDARY OUTCOMES:
Proportion of wounds covered with SSG at 1 week post excision | 1 week
  The proportion of wounds (in percentage) covered with split skin graft at 1 week post excision.
Percentage of graft take at week 1 and week 4 | 4 weeks
  Percentage of skin graft survival at week 1 and week 4
Number of patients with recurrence of HS at 3 and 6 months | 6 months
  Number of patients with recurrence of disease at 3 and 6 months
Number of patients with improved Dermatology Life Quality Index (DLQI) | 6 months
  Dermatology Life Quality Index (DLQI) will be used to measure the improvement in quality of life. Comparison will be made between DLQI during pre operative period and 6 months post operative
The difference in cost between both treatments | 6 months
  Data on the total cost of treatment between both treatment groups will be compared. The total cost will combine the cost of procedures, cost of devices, cost of inpatient stay and cost of clinic follow ups.

CONTACTS AND LOCATIONS:
Overall Officials: Ash Mosahebi, Study Director — Royal Free NHS Foundation Trust London
Locations (1):
- Royal Free NHS Foundation Trust Hospital London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No